CLINICAL TRIAL: NCT02086734
Title: Perfusion CT as a Predictor for Response to Antiangiogenic Therapy in Patients With Metastasized Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Jozefina Casuscelli, Dr. med., Ludwig-Maximilians - University of Munich
Other Study IDs: CTP NK 2012
Record Dates: First submitted 2013-11-28; First posted 2014-03-13 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Renal Cancer
Keywords: Perfusion-CT; mRCC; antiangiogenic therapy; response assessment
MeSH Terms: conditions — Kidney Neoplasms | interventions — Cytidine Triphosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mRCC patients assessed with Perfusion CT: Study population consists of patients with metastasized renal cancer eligible for AAT with either Sunitinib (Sutent®), Pazopanib (Votrient ®), Sorafenib (Nexavar®) evaluated with Perfusion-CT
  Interventions: Other: Perfusion-CT

INTERVENTIONS:
Other: Perfusion-CT — 1. Baseline Perfusion CT-Scan (before AAT)
  2. Follow-Up I Perfusion-CT Scan 7 days after start with AAT
  3. Follow-Up II Perfusion-CT Scan 8 weeks after start with AAT

SUMMARY:
The purpose of this study is the evaluation of dynamic contrast-enhanced CT (Perfusion-CT) for therapeutic response predicition in patients with metastasized renal carcinoma (mRCC) undergoing antiangiogenetic therapy (AAT) with multikinase inhibitors.

In this study patients with mRCC under AAT will be examined with 3 serial Perfusion - CT scans - partially intergrated in their regular staging CT scheme - at baseline (before AAT start), 1 week after AAT as well as 8 weeks after AAT initialization. Thereby selected intrabdomial or intrathoracic metastases will be monitored longitudinally with perfusion CT. Pretreament and post-treament perfusion characteristics of the assessed metastatic lesions will be quantified and correlated with patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients with metastasized renal cell carcinoma treated at the Department of Urology (University of Munich - Grosshadern Campus)

  1. with either - Sunitinib (Sutent®), Pazopanib (Votrient ®) bzw. Sorafenib (Nexavar®) as first-line therapy
  2. with Sunitinib (Sutent®), Pazopanib (Votrient ®) bzw. Sorafenib (Nexavar®) as second-line therapy after failed first-line therapy, who are off therapy for at least 2 weeks
* no contraindications against contrast-enhanced CT
* obtained informed consent to participate in the study

Exclusion Criteria:

Patients who have:

* not given informed consent
* known iodine allergy
* high grade renal insuffiency (eGFR < 30ml/min) not on dialysis
* overt hyperthyreoidism
* singular metastases <1cm in diameter
* an increase of their baseline creatine levels of >20% between CT examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic renal cell cancer eligible for AAT (antiangiogenic therapy) with either Sunitinib (Sutent®), Pazopanib (Votrient ®), Sorafenib (Nexavar®) presenting at the Departement of Urology. LMU, meeting the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Prediction of progression-free interval and overall survival after initialization of antiangiogenic therapy based on baseline values and relative changes of CT perfusion parameters | up to 3 years

SECONDARY OUTCOMES:
Correlation of CT perfusion parameters at baseline as well as their relative changes after start of antiangiogenic therapy with response status according to RECIST 1.1 | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Staehler, Prof. Dr. med., Study Chair — Urologische Klinik und Poliklinik der Universität München; Anno Graser, Prof. Dr. med., Study Director — Institut für Klinische Radiologie des Klinikums der Universität München; Alexander Sterzik, Dr. med., Principal Investigator — Institut für Klinische Radiologie des Klinikums der Universität München; Jozefina Casuscelli, Dr. med., Principal Investigator — Urologische Klinik und Poliklinik der Universität München
Locations (1):
- Urologische Klinik und Poliklinik der Universität München, München, Bavaria, Germany